CLINICAL TRIAL: NCT06923878
Title: Comparison of Prick-to-prick Testing, Extract-specific IgE Antibody Testing and Component Resolved Diagnosis (CRD) in Diagnosing of Allergy to Peas, Lentils, Chickpeas and Green Beans
Brief Title: Comparison of Skin Prick Testing, Extract-specific IgE Antibody Testing and Component Resolved Diagnosis in Diagnosing of Legume Allergy
Acronym: CRD
Status: Recruiting | Type: Observational
Sponsor: University Hospital Pilsen (Other)
Collaborators: MacroArray Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD
Record Dates: First submitted 2025-03-17; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Food Allergy Suspected
Keywords: food allergy; component resolved diagnosis; skin prick test; oral food challenge; legume allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Patients with food allergy
- Group 2: Healthy volunteers

SUMMARY:
The study is aimed at improving the diagnosis of food allergy, specifically allergy to commonly consumed legumes such as peas, lentils, chickpeas or green beans. Patients suspected of allergy to these legumes will be examined using traditional methods of IgE-mediated allergy diagnosing (skin prick test, testing for specific IgE antibodies against food extract), but also by testing for specific IgE antibodies against relevant allergenic molecules of these legumes. The results of performed tests will be compared with the result of the oral food challenge, which is considered to be the gold standard of food allergy diagnosis.

DETAILED DESCRIPTION:
Legumes are one of the major food allergens, but these are usually peanuts or soybeans. Other legumes, such as peas, lentils, chickpeas or green beans, have been overlooked, but some studies suggest that they may also cause allergic reactions ranging from urticaria to anaphylaxis. The prevalence of allergy to these neglected legumes can range widely (0.5-39.6%) depending on the patient group and the method of allergy diagnosis.

The main allergens of legumes are the seed storage proteins, including 7S and 11S globulins and especially 2S albumins, which can cause the most severe, often systemic allergic reactions. These proteins are characterized by their considerable resistance to heat and other physical or chemical influences. Other important legume allergens in our geographical area are the PR-10 proteins cross-reacting with the major allergen of birch pollen (Bet v 1), which in turn are more sensitive to heat treatment and tend to be the source of milder, more local reactions. In contrast, sensitization to other allergen groups, such as lipid transfer proteins (LTPs), oleosins or profilins, is less significant.

ELIGIBILITY:
Inclusion Criteria:

* age: ≤ 65 years
* signing informed consent to the study
* a positive history of an immediate allergic reaction to one or more of the legumes studied (peas, lentils, chickpeas, beans) with skin, gastrointestinal, respiratory or cardiovascular symptoms occurring within 2 hours after ingestion and a positive result of specific IgE testing against ALEX and/or skin prick test with the legume
* patients with a positive OFC with any of the legumes studied

Exclusion Criteria:

* disagreement with the implementation of the oral food challenge
* history of severe systemic allergic reaction to the legume in question (Ring-Messmer grade ≥ 3)

Ages: 4 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: European population, Caucasian race
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Specificity and sensitivity of the tests performed | 6 months
  Specificity and sensitivity of the tests performed

SECONDARY OUTCOMES:
Food challenge protocol | From enrollment and no later than one.
  Food challenge protocol
Specific lultiplex assay including allergenic component of legumes | 6 months
  Specific multiplex assay including legume allergenic components

CONTACTS AND LOCATIONS:
Overall Officials: Martin Liska, MD, Principal Investigator — Department of allergology and immunology
Locations (1):
- University Hospital Pilsen, Pilsen, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Undecided